CLINICAL TRIAL: NCT01130896
Title: Clinically Indicated Magnetic Resonance Imaging of Patients With Permanent Pacemakers (PPM) and Implantable Defibrillators (ICD)
Brief Title: Clinically Indicated Magnetic Resonance Imaging in Patients With Cardiac Devices
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: RPN03-08-12-11
Record Dates: First submitted 2010-05-20; First posted 2010-05-26 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Arrhythmias, Cardiac
Keywords: MRI, pacemakers, Defibrillator
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MRI and Cardiac Devices: Clinically indicated MRI (all types) in patients with implanted pacemakers and ICD

SUMMARY:
Patients with implanted cardiac devices who meet appropriate entrance criteria undergo clinically indicated Magnetic Resonance (MR) Imaging Studies using an established safety protocol.

DETAILED DESCRIPTION:
This prospective cohort study to use an established MRI device safety protocol to decrease the risk of clinically indicated MR imaging in patients with implantable cardiac devices. All devices will undergo a complete interrogation and testing of thresholds, sensing, battery voltage and impedances prior to and following imaging. Pre-MRI, devices will be programmed to setting that will ensure MRI safety. During imaging, patients will blood pressure, heart rate and O2 sat level will be monitored continuously.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an emergent or absolute need for MR imaging and PPM or certain ICD's

Exclusion Criteria:

* Pacemaker dependent patients with ICD's
* Patients with other contraindication to MRI

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Implanted Cardiac Rhythm Management Devices
Sampling Method: Non-Probability Sample
Enrollment: 1509 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry R. Halperin, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Blalcok 5 MRI, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Nazarian S, Hansford R, Rahsepar AA, Weltin V, McVeigh D, Gucuk Ipek E, Kwan A, Berger RD, Calkins H, Lardo AC, Kraut MA, Kamel IR, Zimmerman SL, Halperin HR. Safety of Magnetic Resonance Imaging in Patients with Cardiac Devices. N Engl J Med. 2017 Dec 28;377(26):2555-2564. doi: 10.1056/NEJMoa1604267. PMID 29281579
- [Result] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340
- [Derived] Ra J, Oberdier MT, Suzuki M, Vaidya D, Liu Y, Hansford R, McVeigh D, Weltin V, Tao S, Thiemann DR, Nazarian S, Halperin HR. Implantable Defibrillator System Shock Function, Mortality, and Cause of Death After Magnetic Resonance Imaging. Ann Intern Med. 2023 Mar;176(3):289-297. doi: 10.7326/M22-2653. Epub 2023 Jan 31. PMID 36716451
- [Derived] Rahsepar AA, Zimmerman SL, Hansford R, Guttman MA, Castro V, McVeigh D, Kirsch JE, Halperin HR, Nazarian S. The Relationship between MRI Radiofrequency Energy and Function of Nonconditional Implanted Cardiac Devices: A Prospective Evaluation. Radiology. 2020 May;295(2):307-313. doi: 10.1148/radiol.2020191132. Epub 2020 Mar 3. PMID 32125255
- See also: PubMed Citation #1 — https://pubmed.ncbi.nlm.nih.gov/29281579/
- See also: PubMed Citation #2 — https://pubmed.ncbi.nlm.nih.gov/21969340/

RESULTS

PARTICIPANT FLOW:
Groups:
- MRI and Cardiac Devices: Clinically indicated MRI (all types) in patients with implanted pacemakers and implantable cardioverter-defibrillator (ICD)
Period: Overall Study
Arm/Group | MRI and Cardiac Devices
Started | 1509
Completed | 1509
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | MRI and Cardiac Devices
Number analyzed (Participants) | 1509
Age, Continuous [Mean (Full Range); unit: years] | 69.3 [57.7 to 78.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 548
  Male | 961
Region of Enrollment [Number; unit: participants]
  United States | 1509

OUTCOME MEASURES:

1. Primary Outcome: Device Malfunction
Description: Number of patients with change in device testing defined as a change in any of the following (impedance, battery life, p and r wave sensing and atrial and ventricular capture thresholds) not to exceed 50 percent from baseline
Time Frame: immediately post MRI (up to 2 hours) and long-term follow-up (up to 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Cardiac Devices
Number analyzed (Participants) | 1509
Participants
  immediately post MRI (up to 2 hours) | 24
  Long-term follow-up (up to 6 months) | 52

2. Primary Outcome: Patient Safety
Description: Number of patients with change in vital signs including blood pressure, heart rate and pulse oximetry not to exceed 10 percent from baseline lead impedances as well as patient reports of any discomfort related to MRI)
Time Frame: assessed during MRI and immediate post MRI (up to 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Cardiac Devices
Number analyzed (Participants) | 1509
Participants | 0

3. Secondary Outcome: Noise Artifacts as Assessed by the Number of Participants With a Greater Than a 50% Change in Lead Impedance
Description: We will evaluate whether or not the artifacts produced are significant enough to prevent diagnostic interpretation of images
Time Frame: Immediately post MRI (up to 2 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | MRI and Cardiac Devices
Number analyzed (Participants) | 1509
Participants | 0

ADVERSE EVENTS:
Arm/Group | MRI and Cardiac Devices
All-Cause Mortality (participants affected / at risk) | 0/1509
Serious Adverse Events (participants affected / at risk) | 0/1509
Other Adverse Events (participants affected / at risk) | 8/1509
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MRI and Cardiac Devices (N=1509)
Power on reset (Surgical and medical procedures) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes